CLINICAL TRIAL: NCT04532177
Title: Prospective Pilot Study of Stereotactic Body Radiation Therapy (SBRT) for Invasive Breast Cancer Patients Not Undergoing Definitive Surgery
Brief Title: Stereotactic Body Radiation Therapy (SBRT) for Invasive Breast Cancer Patients Not Undergoing Definitive Surgery
Acronym: SBRT BREAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Alexander Stessin, Clinical Assistant Professor of Medicine, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBU-SBRT-BREAST-NO-SX
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — fractionated linear accelerator based SBRT to 40 Gy in 5 fractions

SUMMARY:
This is a prospective pilot study investigating the safety and efficacy of stereotactic body radiation therapy (SBRT) as a treatment for breast cancer in patients who do not get surgery. The study will accrue 15 patients who will be treated to a dose of 40 Gy over the course of 5 fractions in the Stony Brook University Hospital Department of Radiation Oncology. The subjects will then have a follow up time of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18
* Biopsy proven invasive carcinoma of the breast
* Clinical T1-T4 invasive carcinoma
* Cancer is deemed unresectable with no possibility of future resection or the patient is a poor surgical candidate as determined following evaluation by a surgeon.
* Women who are not post-menopausal should have a negative urine or serum pregnancy test. Women of childbearing potential must agree to adequate contraception for the duration of study participation.
* Ability to understand and willingness to sign a written informed consent document
* Life expectancy > 6 months
* Patient is to be treated at Stony Brook University Hospital

Exclusion Criteria:

* Women with a known pregnancy, positive serum pregnancy test, or currently breastfeeding as well as women of childbearing potential unwilling or unable to use an acceptable method of birth control (including abstinence or barrier method of birth control) to avoid pregnancy for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Breast implant in the breast to be treated with SBRT
* Insufficient breast imaging to judge clinical stage
* Inability to receive study treatment planning and treatment secondary to body habitus
* Inability to understand or unwillingness to sign a written consent document
* Life expectancy < 6 months
* Children (< 18 years of age)
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situation that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Rates of acute and late adverse events grade 3 or greater | 5 years
  Rates of acute and late grade 3 or greater toxicity
Partial and complete response rate by clinical and radiographic response | 5 years

SECONDARY OUTCOMES:
Survival | 5 years
  Progression-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M Stessin, MD, Principal Investigator — Stony Brook Cancer Center
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No